CLINICAL TRIAL: NCT00315718
Title: Controlled Clinical Trial on Long Term Effects of Hintonia Latiflora Extract in Mild to Moderate Type 2 Diabetes
Brief Title: Long-Term Effects of Sucontral(TM) on Mild and Moderate Cases of Diabetes Mellitus (Type 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harras Pharma Curarina GmbH (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPC-02/1998
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2006-04-19 (Estimated); Status verified 2006-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Hintonia latiflora extract; Diabetes mellitus type 2; HbA1c; Safety; Liver function tests
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Extract from Hintonia latiflora bark

SUMMARY:
In patients with diabetes mellitus type 2 stably adjusted to diet long-term intake of aqueous-ethanolic extract from Hintonia latiflora over more than 12 months leads to a statstically significant amelioration of parameters of glycaemic control (HbA1c, postprandial and fasting glucose) not acchievable with diet alone.

As safety parameters, liver function tests and cardiovascular parameters are to be monitored. Adverse events are to be monitored.

DETAILED DESCRIPTION:
Objective:

To evaluate the long term effects of an aqueous-ethanolic extract from the bark of Hintonia latiflora (1:4.5, extraction medium 32% ethanol) in mild to moderate cases of type II diabetes, especially on parameters of glycaemic control and safety.

Research Design and Methods:

The trial was carried out as a controlled single-centre open study. 30 patients stably adjusted to diet were treated with the study medication (3 x 2 ml/day before meals) for up to 36 months. Efficacy parameters were HbA1c and fasting and postprandial serum glucose. As parameters for safety, liver function tests, cardiac functions and adverse events were assessed.

Results:

All three efficacy parameters improved significantly, and the parameters of glycaemic control remained stable for the study duration of 36 months. As compared to baseline, after 6 months and 18 months of therapy mean fasting glucose was reduced by 23.9 and 21.9 % (1.8 mmol and 2.0 mmol in absolute values). Mean postprandial glucose was reduced by 24.4 and 16.5 % (2.4 and 2.0 mmol in absolute values), and the mean HbA1c was decreased by 10.4 and 12.4 % (0.76 and 1.04% in absolute figures). Improvement was maintained after 18 months. Tolerability was excellent. No hypoglycaemic reactions occurred. No adverse effects or change in cardiac and liver function tests were observed. There was a tendency towards decreasing triglyceride and total cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Diabetes mellitus type 2 stable adjusted to diet
* Minimum duration of diabetic complaints 1 year
* Fasting serum glucose 7-14 mmol/l
* HbA1c max. 12%
* Written consent

Exclusion Criteria:

* Hepatic impairment
* Renal impairment
* Pregnancy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2002-06; Study Completion 2005-06

PRIMARY OUTCOMES:
HbA1c values

SECONDARY OUTCOMES:
Postprandial blood glucose
Fasting blood glucose
General vegetative symptoms
BMI
Liver function tests (ALT, GGT, AP)
Serum lipids (triglycerides, cholesterol, HDL cholesterol)
Adverse drug reactions (narratives)
Blood pressure (systolic/diastolic)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Korecova, Dr. med., Principal Investigator — Head of Diabetes Department, IDF President, Rc: 425201/734, Vel'komoravská 2, SK-91101 Trencin
Locations (1):
- Hospital of Trencin, Trenčín, Slovakia